CLINICAL TRIAL: NCT02695771
Title: A Prospective, Open-label Randomized Clinical Trial of a Single Bladder Instillation of Mitomycin C vs. Gemcitabine vs. No Additional Treatment Immediately After Transurethral Resection of Bladder Tumor (TURBT)
Brief Title: The Bladder Instillation Comparison Study
Acronym: BIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Brian R. Lane, Urologist, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-030
Record Dates: First submitted 2016-02-09; First posted 2016-03-01 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Urinary Bladder Neoplasms
Keywords: bladder tumors; urinary tumors; non-muscle invasive bladder tumors; NMIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mitomycin C (Experimental): Mitomycin C 40 mg in 40 mL of 0.9% sodium chloride intravesicular immediately following TURBT one time.
  Interventions: Drug: Mitomycin C
- Gemcitabine (Active Comparator): Gemcitabine 2 grams in 100 mL of 0.9% sodium chloride intravesicular immediately following TURBT one time.
  Interventions: Drug: Gemcitabine
- No intervention (No Intervention): Patients randomized to this arm will receive no intervention intravesicular immediately following TURBT one time.

INTERVENTIONS:
Drug: Mitomycin C — Cancer chemotherapeutic agent
  Other Names: Mutamycin
  Arms: Mitomycin C
Drug: Gemcitabine — Cancer chemotherapeutic agent
  Other Names: Gemzar, Novaplus
  Arms: Gemcitabine

SUMMARY:
To compare the efficacy of Mitomycin C vs. Gemcitabine vs. no adjuvant treatment as a single intraoperative instillation in preventing recurrence of bladder cancer.

DETAILED DESCRIPTION:
This study will compare standard of care treatment for patients with non-muscle invasive bladder cancer (NMIBC). Patients will be randomized to one of three arms, Mitomycin C, Gemcitabine or no additional treatment immediately following TURBT in the operating suite. All treatment, surgical procedures and follow up care will be conducted according to standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. sign an informed consent for the study
2. be scheduled for a TURBT for suspected non-muscle invasive bladder tumor.

Exclusion Criteria:

1. patients unable to consent for themselves
2. individuals under 18 years old
3. pregnant women
4. prisoners
5. patients with known allergy or intolerance to the mitomycin C or Gemcitabine
6. any other sound medical, psychiatric and/or social reason as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Lane, MD, Principal Investigator — Corewell Health West
Locations (3):
- United States (3):
  - Spectrum Health Medical Group-Division of Urology-LHCP, Grand Rapids, Michigan
  - Spectrum Health Medical Group-Division of Urology, Grand Rapids, Michigan
  - Urologic Consultants P.C., Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weijers Y, Arentsen HC, Arends TJ, Witjes JA. Management of low-risk and intermediate-risk non-muscle-invasive bladder carcinoma. Hematol Oncol Clin North Am. 2015 Apr;29(2):219-25, vii. doi: 10.1016/j.hoc.2014.11.001. PMID 25836930
- [Background] Pagano MJ, Badalato G, McKiernan JM. Optimal treatment of non-muscle invasive urothelial carcinoma including perioperative management revisited. Curr Urol Rep. 2014 Nov;15(11):450. doi: 10.1007/s11934-014-0450-1. PMID 25234184
- [Background] Roupret M, Babjuk M, Comperat E, Zigeuner R, Sylvester RJ, Burger M, Cowan NC, Bohle A, Van Rhijn BW, Kaasinen E, Palou J, Shariat SF. European Association of Urology Guidelines on Upper Urinary Tract Urothelial Cell Carcinoma: 2015 Update. Eur Urol. 2015 Nov;68(5):868-79. doi: 10.1016/j.eururo.2015.06.044. Epub 2015 Jul 16. PMID 26188393
- [Background] Sylvester RJ, Oosterlinck W, van der Meijden AP. A single immediate postoperative instillation of chemotherapy decreases the risk of recurrence in patients with stage Ta T1 bladder cancer: a meta-analysis of published results of randomized clinical trials. J Urol. 2004 Jun;171(6 Pt 1):2186-90, quiz 2435. doi: 10.1097/01.ju.0000125486.92260.b2. PMID 15126782
- [Background] Au JL, Badalament RA, Wientjes MG, Young DC, Warner JA, Venema PL, Pollifrone DL, Harbrecht JD, Chin JL, Lerner SP, Miles BJ; International Mitomycin C Consortium. Methods to improve efficacy of intravesical mitomycin C: results of a randomized phase III trial. J Natl Cancer Inst. 2001 Apr 18;93(8):597-604. doi: 10.1093/jnci/93.8.597. PMID 11309436
- [Background] Montgomery JS, Miller DC, Weizer AZ. Quality indicators in the management of bladder cancer. J Natl Compr Canc Netw. 2013 Apr 1;11(4):492-500. doi: 10.6004/jnccn.2013.0061. PMID 23584349
- [Derived] Han MA, Maisch P, Jung JH, Hwang JE, Narayan V, Cleves A, Hwang EC, Dahm P. Intravesical gemcitabine for non-muscle invasive bladder cancer. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD009294. doi: 10.1002/14651858.CD009294.pub3. PMID 34125951

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: recruitment goals were not met as study was stopped early by the IRB. Enrollment was suspended due to protocol deviations concerning randomization and physician bias.
Period: Overall Study
Arm/Group | Mitomycin C | Gemcitabine | No Intervention
Started | 29 | 26 | 27
Completed | 29 | 26 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitomycin C | Gemcitabine | No Intervention | Total
Number analyzed (Participants) | 29 | 26 | 27 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 8 | 22
  >=65 years | 23 | 18 | 19 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74 [66 to 80] | 69 [61 to 81] | 74 [62 to 81] | 73 [64 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 15
  Male | 24 | 22 | 21 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 28 | 24 | 25 | 77
  African American | 0 | 2 | 1 | 3
  Refused to answer | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 26 | 27 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Grade ≥ 3 Adverse Event, Graded According to NCI CTCAE Version 4.03
Description: The NCI CTCAE Version 4.03 grades adverse events as follows: grade 3 include severe but non-life-threatening consequences that result in hospitalization and/or interventions, including elective radiologic or operative interventions; grade 4 events include life-threatening consequences, such as those requiring urgent reoperation; and grade 5 events result in treatment-related death.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | Mitomycin C | Gemcitabine | No Intervention
Number analyzed (Participants) | 29 | 26 | 27
Participants | 15 | 14 | 20

2. Secondary Outcome: Freedom From Bladder Stones/Dystrophic Calcification
Description: The secondary endpoint for this study will be the number of subjects who did not experience dystrophic calcification or bladder calculi measured by the number of patients with Grade 3 through Grade 5 Adverse Events that are related to study arm, graded according to NCI CTCAE Version 4.03.Version 4.03
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | Mitomycin C | Gemcitabine | No Intervention
Number analyzed (Participants) | 29 | 26 | 27
Participants | 24 | 23 | 25

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Mitomycin C | Gemcitabine | No Intervention
All-Cause Mortality (participants affected / at risk) | 2/29 | 1/26 | 1/27
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/26 | 1/27
Other Adverse Events (participants affected / at risk) | 9/29 | 5/26 | 5/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitomycin C (N=29) | Gemcitabine (N=26) | No Intervention (N=27)
Femoral Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — Right subcapital femoral neck fracture and patient was admitted to orthopedic surgery.
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 — Persistent hematuria with clot retention requiring foley catheter and continuous bladder irrigation. Patient underwent cystoscopy with clot evacuation and fulguration
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 — cardiac arrest secondary to ventricular fibrillation with inferior STEMI
Thromboembolic Event (Blood and lymphatic system disorders) | 0 | 0 | 1 — Left lower extremity claudication with history of left superficial femoral artery stent with thrombosis of stent
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitomycin C (N=29) | Gemcitabine (N=26) | No Intervention (N=27)
Dystrophic calcification/bladder stone (Renal and urinary disorders) | 5 (11) | 3 (8) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Fever (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The limitations of this study are evident given the early closure and being underpowered. Enrollment was suspended due to protocol deviations concerning randomization and physician bias. A review of the protocol deviations revealed the primary errors made were noted during the consent process. Specifically, patients were consented by individuals not identified as part of the research team and others consented the day of the procedure, both in violation of the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT02695771/Prot_SAP_000.pdf